CLINICAL TRIAL: NCT01225692
Title: Brain Trauma Outcomes in Nova Scotia
Brief Title: Brain Trauma Outcomes in Nova Scotia Study
Acronym: BTOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Dr. B. David Clarke, QEII HSC,Capital Health, Dalhousie University, Division of Neursosurgery
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: CDHA-RS/2004-014; PSO-Project- 2003-353 (Other Grant/Funding Number: Nova Scotia Health Research Foundation)
Record Dates: First submitted 2010-10-15; First posted 2010-10-21 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Brain Injuries,Traumatic; Outcome Assessment (Health Care); Craniocerebral Trauma; Emergency Medical Services; Organizational Innovation
Keywords: Brain Injury; Head Trauma; Trauma Systems; Head Injury Guideline; Time to Tertiary Care
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Head Injury Guideline

SUMMARY:
The goals of this study are to identify outcome indicators of optimal care for brain injury patients, including pre-hospital care, prompt delivery to neurosurgical care and access to early rehabilitation services. Nova Scotia's centralized Neurosurgical services and integrated provincial Emergency Health Services provide a rich opportunity to construct a cohesive, integrated data management system. This system will allow us to answer important research questions related to the outcomes, care and prevention of brain trauma.

Retrospective data collection The retrospective arm of the BTO study has created full data sets and care pathways from multiple sources covering the continuum of brain trauma care. Investigators continue to analyze this large amount of data and prepare it for publication.

Prospective data Collection Patients with a major head injury (initial GCS 3-12), have been considered for enrollment in the BTO study.The prospective arm of the BTO study has 52 patients enrolled. Screening and Enrollment was complete on June 30, 2007. These patients are participating in long term follow up at 6, 12 and 24 months post injury for assessment of qualitative and quantitative outcomes. Completion of patient follow up will be in June 2009.

ELIGIBILITY:
Retrospective Arm Cohort 1: AIS ≥ 3, head +/- other injuries Cohort 2: AIS ≥ 3, isolated head injury (cohort 2 is a subset of cohort 1)

Inclusion Criteria:

1.patient treated in at least one facility prior to arrival at QEII.

Exclusion Criteria

1. injured out of province
2. time from injury to 1st facility presentation known to be > 24 hours
3. time arrival at 1st referring facility to time arrive at QEII known to be > 24 hours
4. direct ground or air scene transport

Prospective Arm:

Inclusion Criteria:

1. have a head injury requiring hospital admission
2. able to provide informed consent or have next- of -kin able to provide consent on patients' behalf

Exclusion Criteria:

1. unwilling or unable to provide consent

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-02; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Time Measurement; Hours:minutes
  Time as measured by ; Time Elapsed from Injury Time to Time of Arrival at Tertiary Care

SECONDARY OUTCOMES:
Clinical Follow-up; Numerical Score 1-5;Glasgow Outcome Scores (GOS)
  Glasgow Outcome Scores (GOS)
  Score ranges from:
  5 Good Recovery (Resumption of normal life despite minor deficits) 4 Moderate Disability(Disabled but independent. Can work in sheltered setting) 3 Severe Disability (Conscious but disabled. Dependent for daily support) 2 Persistent vegetative (Minimal responsiveness)
  1 Death (Non survival)